CLINICAL TRIAL: NCT01866098
Title: Naltrexone for Antipsychotic-Induced Weight Gain
Acronym: NTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1207010507; 1R01DK093924-01A1 (NIH)
Record Dates: First submitted 2013-03-12; First posted 2013-05-31 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Bipolar Disorder; Severe Major Depression With Psychotic Features
Keywords: antipsychotic; severe mental illness; weight loss
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Mental Disorders; Weight Loss | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Naltrexone 50mg (Experimental): Oral Naltrexone 50mg capsule taken once daily for 52 weeks
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Oral placebo capsule taken once daily for 52 weeks
  Interventions: Drug: Placebo
- Naltrexone 25mg (Experimental): Oral Naltrexone 25mg capsule taken once daily for 52 weeks
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — 25 or 50mg (randomized) oral capsule taken once daily for 52 weeks to establish optimal dose for weight loss over the course of the study.
  Other Names: Revia
  Arms: Naltrexone 25mg; Naltrexone 50mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to look at the effects of naltrexone on weight loss in individuals treated with antipsychotic medications. Naltrexone is an FDA approved medication for the management of alcohol dependence and drug dependence, but has not been fully evaluated for its effect on weight loss in individuals with severe mental illness (i.e. schizophrenia, schizoaffective disorder, bipolar disorder etc.) The purpose of this study is to find out how effective two different doses of oral naltrexone is on reducing body weight when compared to placebo (an inactive substance or "sugar pill").

DETAILED DESCRIPTION:
Persons with severe mental illness (SMI) die, on average, 25 years earlier than the general population1. Most of this early mortality can be attributed to cardiovascular disease (CVD) and diabetes mellitus (DM), which are directly related to obesity. Obesity is a leading cause of preventable death in the United States, second only to smoking. The physical health of patients has become a major focus of schizophrenia care, as recent decades have seen immense gains in symptom control and community integration. There is an urgent need for the development of interventions that address the obesity crisis in schizophrenia.

Patients treated with antipsychotic medications have been shown to have a preference for diets high in fat and sugar. Patients with schizophrenia typically seek behaviors that increase dopamine mediated reward in the brain such as smoking and substance use, both of which occur more often in this group than the general population. The system might require intact dopamine and opioid function.

Naltrexone is an oral agent that competitively antagonizes all known opioid receptors in the brain. Human studies with naltrexone were completed in individuals with different illnesses, including schizophrenia, and have been shown to be a safe and easy agent to use. It is shown to decrease craving in alcoholics and is approved by the FDA for the treatment of alcohol dependence. Naltrexone is reported to decrease craving for other substances of abuse, like nicotine. Furthermore, it has been shown to prevent secondary weight gain due to cessation of cigarette smoking at low (25mg and 50 mg), but not higher doses. Naltrexone has been tested in human feeding studies, and has been shown to reduce both the quantity of food eaten and the choice of palatable foods.

Subjects will be randomized to either 25, 50 or 0mg of Naltrexone and will take the study medication daily for 52 weeks. Subjects will be seen weekly for the first 4 weeks of the study, thereafter they will be seen on a bi-weekly (every other week) basis to be assessed (i.e. weight, side effect check, paper questionnaires) throughout the remaining 48 weeks of treatment.

The purpose of this study is to determine the efficacy of two doses of naltrexone (25mg & 50mg) versus placebo for weight and health risk reduction in 144 obese individuals with severe mental illness treated with an antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75
* Meet Diagnostic & Statistical Manual - 4 (DSM-IV) criteria for schizophrenia, schizoaffective disorder, bipolar disorder, major depression, or another psychotic disorder based on Structured Clinical Interview for the DSM-IV (SCID) interview
* Body Mass Index (BMI) of 28 and over
* On a stable dose of antipsychotic medication; i.e. at least one month with no dose change, and three months from an antipsychotic switch
* Deemed to be symptomatically stable by the clinical staff in the last two months
* Over 7% total body weight increase on antipsychotics for subjects within first year of illness

Exclusion Criteria:

* Meet criteria for current opiate abuse or dependence (confirmed by positive urine drug screen for opiates or, if suspected by study doctor via patient history and or suspicion of occult opiate use, a naloxone challenge will be performed.)
* Current history of dementia, mental retardation
* Not capable of giving informed consent for participation in the study
* Women who are pregnant or breast-feeding
* Physical conditions affecting body weight (e.g. Cushing's disease, polycystic ovary syndrome) Diabetes Mellitus (defined as prescribed an anti-diabetic medication for diabetes or a hemoglobin A1c level > 7 confirmed by primary care physician at screening)
* Severe liver dysfunction, (serum aminotransferases greater than three times normal), acute infectious hepatitis, liver failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-05; Primary Completion 2019-04-07 (Actual); Study Completion 2019-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data resulting from this award involving human subjects will be submitted to the NIMH Data Archive (NDA) - National Database for Clinical Trials Related to Mental Illness (NDCT) The Principal Investigator will work with NDA support staff to plan an appropriate data submission schedule and provide information on the steps for submission and sharing of data. Communication of this data sharing plan to appropriate research staff to ensure the timely submission of data. All human subject data provided will include an NDA Global Unique Identifier (GUID) and will not include personally identifiable information (PII). Analyzed data will be submitted no later than the time of publication. Even if a publication focuses on only part of an analyzed dataset, the entire analyzed dataset will be submitted when the first paper is published. All data made available for public use via NDA will be de-identified data.

REFERENCES:
- [Derived] Tek C, Guloksuz S, Srihari VH, Reutenauer EL. Investigating the safety and efficacy of naltrexone for anti-psychotic induced weight gain in severe mental illness: study protocol of a double-blind, randomized, placebo-controlled trial. BMC Psychiatry. 2013 Jun 27;13:176. doi: 10.1186/1471-244X-13-176. PMID 23805859

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral placebo capsule taken once daily for 52 weeks
  Placebo
Period: Overall Study
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Started | 51 | 47 | 46
Completed | 32 | 20 | 25
Not Completed | 19 | 27 | 21
Not completed — Lost to Follow-up | 11 | 18 | 13
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Adverse Event | 1 | 5 | 4
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Unrelated Hospitalization | 2 | 0 | 1
Not completed — Non-compliance | 1 | 0 | 1
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg | Total
Number analyzed (Participants) | 51 | 47 | 46 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.8) | 45.0 (11.5) | 43.0 (14.2) | 43.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 25 | 77
  Male | 21 | 25 | 21 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 18 | 16 | 27 | 61
  African American | 24 | 28 | 16 | 68
  Other | 9 | 3 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United States | 51 | 47 | 46 | 144
Body Mass Index (BMI) [Mean (Standard Deviation); unit: weight in kg/ height m^2] — BMI = weight in kg/ height m^2
  weight in kg/ height m^2 | 39.1 (7.3) | 37.1 (5.7) | 38.9 (11.4) | 38.4 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline
Description: Weight (kilograms; kg) will be measured at each assessment and change in weight will be determined at study endpoint.
Time Frame: Baseline and 52 weeks
Population: Analysis population consists of participants who were randomized, received at least 1 dose of the trial compound (naltrexone or placebo), and had at least 1 assessment after baseline.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
kg | -0.16 (1.78) | 0.69 (2.22) | -0.95 (2.06)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.83, Mixed Models Analysis; Estimated treatment differences between groups analyzed using mixed-model analysis. Model includes the baseline value age; sex; compliance; ethnicity

2. Primary Outcome: Percent of Subjects Who Lost More Than 5% of Body Weight From Baseline
Description: Body Mass Index will be calculated at each assessment and change over time will be assessed at endpoint.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
Participants | 10 | 4 | 9
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.10, Chi-squared

3. Secondary Outcome: Changes in Fasting Glucose From Baseline
Description: Fasting glucose will be collected over the course of participation and changes will be evaluated at study endpoint.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
mg/dL | 8.2 (2.6) | 4.6 (3.2) | -0.4 (2.9)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.19, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Changes in Glycosylated Hemoglobin (HbA1c) From Baseline
Description: Glycosylated hemoglobin (HbA1c) will be collected over the course of participation and changes will be evaluated at study endpoint.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
mg/dL | -0.007 (0.11) | -0.061 (0.15) | 0.060 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.96, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Changes in Insulin From Baseline
Description: Insulin will be collected over the course of participation and changes will be evaluated at study endpoint.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
mg/dL | 6.45 (4.89) | 0.45 (6.23) | 2.16 (5.55)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.92, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Changes in Total Cholesterol From Baseline
Description: Total Cholesterol will be collected over the course of participation and changes will be evaluated at study endpoint.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
mg/dL | -1.16 (5.12) | 1.52 (6.41) | -3.02 (5.72)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg; Test type: Superiority; p = 0.98, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Changes in HDL From Baseline
Description: High-density lipoprotein (HDL) will be collected over the course of participation and changes will be evaluated at study endpoint.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
mg/dL | 0.04 (1.73) | 0.79 (2.19) | 0.36 (1.93)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.95, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Changes in LDL From Baseline
Description: Low-density lipoprotein (HDL) will be collected over the course of participation and changes will be evaluated at study endpoint.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
Number analyzed (Participants) | 51 | 47 | 46
mg/dL | -10.87 (4.47) | 1.14 (5.46) | -4.40 (4.91)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 25mg vs Naltrexone 50mg; Test type: Superiority; p = 0.43, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 52 weeks.
Arm/Group | Placebo | Naltrexone 25mg | Naltrexone 50mg
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/47 | 0/46
Other Adverse Events (participants affected / at risk) | 35/51 | 33/47 | 35/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Naltrexone 25mg (N=47) | Naltrexone 50mg (N=46)
Cocaine Overdose (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Naltrexone 25mg (N=47) | Naltrexone 50mg (N=46)
Concentration difficulties (Nervous system disorders) | 0 | 0 | 3
Asthenia/Fatigability (General disorders) | 2 | 2 | 5
Sleepiness/Sedation (Nervous system disorders) | 3 | 5 | 2
Depression (Psychiatric disorders) | 3 | 2 | 0
Tension/Inner unrest (General disorders) | 1 | 3 | 1
Increased sleep (Nervous system disorders) | 3 | 5 | 1
Reduced sleep (Nervous system disorders) | 7 | 3 | 10
Headache (Nervous system disorders) | 15 | 11 | 13
Reduced salivation (Gastrointestinal disorders) | 6 | 1 | 1
Nausea (Gastrointestinal disorders) | 21 | 20 | 19
Diarrhea (Gastrointestinal disorders) | 11 | 6 | 7
Constipation (Gastrointestinal disorders) | 11 | 10 | 7
Dizziness (Nervous system disorders) | 8 | 8 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Diminished sexual desire (Psychiatric disorders) | 1 | 2 | 3
Stomach pain (Gastrointestinal disorders) | 0 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT01866098/Prot_SAP_000.pdf